CLINICAL TRIAL: NCT07266181
Title: Safety and Efficacy of CD19 Chimeric Antigen Receptor T-Cell Immunotherapy (CAR-T) in the Treatment of Refractory Membranous Nephropathy
Brief Title: Safety and Efficacy of CD19 Chimeric Antigen Receptor T-Cell (CAR-T) in the Treatment of Refractory Membranous Nephropathy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Air Force Medicial University (Other)
Responsible Party: Principal Investigator, Li Jipeng, Research associate, The First Affiliated Hospital of Air Force Medicial University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20252388-F-1
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08

CONDITIONS: Refractory Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- To preliminarily evaluate the safety and efficacy of CD19 CAR-T in refractory membranous nephropathy (Other)
  Interventions: Other: All patients will receive CD19 CAR-T cell therapy on the basis of standard symptomatic and supportive treatment.

INTERVENTIONS:
Other: All patients will receive CD19 CAR-T cell therapy on the basis of standard symptomatic and supportive treatment. — Prior to receiving CAR-T cell therapy, patients will undergo lymphodepletion chemotherapy with cyclophosphamide (fludarabine will be added if necessary). After prophylactic administration of antihistamines and acetaminophen, patients will be infused with CD19 CAR-T cells at a dose of 1×10⁶ cells/kg.

SUMMARY:
This study is a single-center, prospective, exploratory Phase I clinical trial initiated by the team led by Associate Professor He Lijie from the Department of Nephrology, Xijing Hospital.

Prior to receiving CAR-T cell therapy, patients will undergo lymphodepletion chemotherapy with cyclophosphamide (fludarabine will be added if necessary). After prophylactic administration of antihistamines and acetaminophen, patients will be infused with CD19 CAR-T cells at a dose of 1×10⁶ cells/kg.

In the subsequent 2 weeks, patients will be hospitalized for monitoring of vital signs and adverse reactions. The planned follow-up duration of this study is 1 years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed as primary membranous nephropathy (PMN) by renal biopsy.
* Classified as moderate-risk or high-risk refractory membranous nephropathy (rMN).
* Moderate-risk rMN is defined as: eGFR ≥ 90 ml/min/1.73m² AND 24-hour urinary protein > 3.5g/d, with a reduction of no more than 50% within 6 months of receiving renin-angiotensin system inhibitor (RASi) therapy.
* High-risk rMN is defined as meeting one of the following:

  1. eGFR < 60 ml/min/1.73m² and/or persistent proteinuria > 8g/d for more than 6 months.
  2. Normal eGFR with proteinuria > 3.5g/d and ≤50% reduction after 6 months of RASi therapy, PLUS at least one of the following: Serum albumin < 25g/L; PLA2R antibody > 50 RU/mL; Urinary α1-microglobulin > 40 μg/min; Urinary IgG > 1 μg/min; Urinary β2-microglobulin > 250 mg/d; IgG/albumin clearance ratio > 0.20.
* Diagnosis of rMN requires failure of adequate first-line immunosuppressive therapy (≥6 months of steroids+cyclophosphamide, CNI, or rituximab), defined by any of the following: persistent high-titer anti-PLA2R antibody; for antibody-negative patients, persistent nephrotic syndrome (protein >3.5g/d, albumin <30g/L); <50% reduction in proteinuria.
* Age ≥ 18 years.
* Adequate organ function, defined as:

  1. Renal: eGFR ≥ 30 ml/min/1.73m².
  2. Hepatic: ALT and AST ≤ 2.5 x ULN; Total bilirubin ≤ 1.5 x ULN.
  3. Cardiac: LVEF ≥ 50%; NYHA Class I or II; No significant arrhythmias requiring intervention; No major cardiovascular events within the past 6 months.
  4. Respiratory: SpO2 > 92% on room air.
* Ability to understand and willingness to sign an Informed Consent Form.

Exclusion Criteria:

* Secondary membranous nephropathy (e.g., due to SLE, malignancy, drugs, infection).
* Active infection requiring IV antibiotics, active tuberculosis, or positive viral serology indicating active infection, including:

  1. HBV: HBsAg (+) and/or HBcAb (+) with detectable HBV DNA.
  2. HCV: HCV Ab (+) with detectable HCV RNA.
  3. HIV Ab (+).
  4. Active EBV or CMV infection (IgM+ or DNA above normal).
  5. Positive syphilis (Treponema pallidum) antibody (requires evaluation for active infection).
* Severe uncontrolled comorbidities, including:

  1. Uncontrolled hypertension (persistent SBP > 160 mmHg or DBP > 100 mmHg).
  2. Uncontrolled diabetes (HbA1c > 8% or random glucose ≥11.1 mmol/L) or diabetic nephropathy.
  3. Symptomatic deep vein thrombosis or pulmonary embolism within the past 6 months.
  4. Active peptic ulcer or gastrointestinal bleeding within the past 6 months.
  5. Severe congenital or acquired immunodeficiency.
  6. Severe CNS diseases (e.g., catastrophic APS, uncontrolled epilepsy).
  7. End-stage organ failure not attributable to PMN.
* History of malignancy within the past 5 years, except for adequately treated non-melanoma skin cancer, cervical carcinoma in situ, or thyroid cancer.
* Specific treatment history or plans, including:

  1. Prior receipt of any cell therapy (e.g., MSCs, HSCT).
  2. Major surgery within 24 weeks before or planned within 24 weeks after enrollment.
  3. Planned kidney transplantation within 3 years.
  4. History of substance abuse.
* Participation in another interventional clinical trial within 3 months prior to enrollment.
* Pregnant or lactating women.
* Inability to understand the study or provide informed consent (e.g., severe dementia, mental illness).
* Any other condition deemed by the investigator to increase risk, interfere with assessment, or affect compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT in rMN subjects after a single infusion of CD19 CAR-T cells | 28 days and 3 months after infusion
  Definition: The DLT evaluated in this study is assessed within two time windows: 28 days (Day 0 to Day 28) and 3 months (Day 28 to Month 3) after CAR-T cell infusion. These time windows are selected based on the typical timeline of CAR-T cell expansion, activity, and potential occurrence of major toxicities in vivo.
  The determination of DLT must meet all the following criteria:1.DLT must be an adverse event judged by the investigator as probably or definitely related to CAR-T cell infusion, and cannot be attributed to underlying diseases, comorbidities, or toxicities from concomitant medications;2.The adverse event must reach a severity grade of ≥ Grade 3 (per CTCAE v5.0) or ≥ Grade 3 specific toxicity grading criteria (e.g., IEC-HS grading).
Incidence of AE in rMN subjects after a single infusion of CD19 CAR-T cells | 12 months after infusion
  Severity grading is based on the Common Terminology Criteria for Adverse Events (CTCAE) v5.0:
  Grade 1: Mild; asymptomatic or mild symptoms; only clinically or diagnostically detectable; no treatment required.
  Grade 2: Moderate; requires minor, local, or non-invasive treatment; limitation in age-appropriate instrumental activities of daily living.
  Grade 3: Severe or medically significant but not immediately life-threatening; results in hospitalization or prolongation of existing hospitalization; disabling; limitation in self-care activities of daily living.
  Grade 4: Life-threatening; requires urgent treatment. Grade 5: Death related to complications.

SECONDARY OUTCOMES:
Overall response rate (CR+PR) in rMN subjects after cell infusion | Week 2, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18 (if applicable), Month 24 (if applicable) after infusion
  1. Definition of rMN CR: Disappearance of the patient's clinical symptoms and signs; urine protein reduced to <0.3 g/day or UACR <300 mg/g; with normal levels of serum albumin (ALB) and serum creatinine (Scr).
  2. Definition of rMN PR: Improvement in clinical symptoms and signs; urine protein decreased by more than 50% compared with baseline, and reduced to 0.3-3.5 g/day or UACR 300-3500 mg/g.
Proportion of rMN subjects achieving CR after cell infusion | Week 2, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18 (if applicable), Month 24 (if applicable) after infusion
  Definition of rMN CR: Disappearance of the patient's clinical symptoms and signs; urine protein reduced to <0.3 g/day or UACR <300 mg/g; with normal levels of serum albumin (ALB) and serum creatinine (Scr).
Proportion of rMN subjects achieving PR after cell infusion | Week 2, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18 (if applicable), Month 24 (if applicable) after infusion
  Definition of rMN PR: Improvement in clinical symptoms and signs; urine protein decreased by more than 50% compared with baseline, and reduced to 0.3-3.5 g/day or UACR 300-3500 mg/g.
rMN recurrence after cell infusion | Week 2, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18 (if applicable), Month 24 (if applicable) after infusion
  Definition of rMN recurrence: After NR or PR, the patient's urine protein rises again to >3.5 g/day or UACR >3500 mg/g; frequent recurrence is defined as more than 2 recurrences within 6 months or more than 4 recurrences within 12 months.
eGFR | Week 2, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18 (if applicable), Month 24 (if applicable) after infusion
  Change in eGFR from baseline in rMN subjects after a single infusion of CD19 CAR-T cells. Estimated glomerular filtration rate, calculated using the CKD-EPI 2021 formula
Urine protein | Week 2, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18 (if applicable), Month 24 (if applicable) after infusion
  Change in urine protein from baseline in rMN subjects after a single infusion of CD19 CAR-T cells, 24-hour urine protein quantification
UACR | Week 2, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18 (if applicable), Month 24 (if applicable) after infusion
  Change in UACR from baseline in rMN subjects after a single infusion of CD19 CAR-T cells, Random urine
anti-PLA2R antibody | Week 2, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18 (if applicable), Month 24 (if applicable) after infusion
  Change in serum anti-PLA2R antibody from baseline in rMN subjects after a single infusion of CD19 CAR-T cells. Venous blood
Scr, CysC | Week 2, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18 (if applicable), Month 24 (if applicable) after infusion
  Change in serum renal function from baseline in rMN subjects after a single infusion of CD19 CAR-T cells.Venous blood
Routine blood test | Week 2, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18 (if applicable), Month 24 (if applicable) after infusion
  Change in blood cells in rMN subjects after a single infusion of CD19 CAR-T cells.Venous blood
CRP | Day 2, Day 7, Day 10 or 14, Day 21, Day 28 (1 month) after infusion
  Change in CRP in rMN subjects after a single infusion of CD19 CAR-T cells.Venous blood
Serum complements C3, C4 | Week 2, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18 (if applicable), Month 24 (if applicable) after infusion
  Change in complements in rMN subjects after a single infusion of CD19 CAR-T cells.
IgE、IgA、IgG、IgM | Week 2, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18 (if applicable), Month 24 (if applicable) after infusion
  Change in immunoglobulins in rMN subjects after a single infusion of CD19 CAR-T cells.
CAR copy number | Day 2, Day 5, Day 7, Day 10 or 14, Day 21, Day 28 (1 month), Month 2, Month 3, Month 6, Month 9, Month 12, Month 18 (if applicable), Month 24 (if applicable) after infusion
  Change in CAR copy parameters in rMN subjects after a single infusion of CD19 CAR-T cells
Ferritin level | Day 2, Day 7, Day 10 or 14, Day 21, Day 28 (1 month) after infusion
  Change in ferritin in rMN subjects after a single infusion of CD19 CAR-T cells
Cytokine panel | Day 2, Day 7, Day 10 or 14, Day 21, Day 28 (1 month) after infusion
  Change in cytokines in rMN subjects after a single infusion of CD19 CAR-T cells
Peripheral blood lymphocyte subset count | Day 2, Day 5, Day 7, Day 10 or 14, Day 21, Day 28 (1 month) after infusion
  Change in peripheral blood lymphocyte subsets in rMN subjects after a single infusion of CD19 CAR-T cells
The surface of peripheral blood B cell subsets | Day 2, Day 5, Day 7, Day 10 or 14, Day 21, Day 28 (1 month) after infusion
  Expression level of CD19 on the surface of peripheral blood B cell subsets in rMN subjects after a single infusion of CD19 CAR-T cells

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology, Xijing Hospital, Xi'an, China, China

DOCUMENTS (4):
  • Study Protocol: English Translation Version (2025-10-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT07266181/Prot_000.pdf
  • Study Protocol: in Simplified Chinese (2025-10-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT07266181/Prot_001.pdf
  • Informed Consent Form: English Translation Version (2025-10-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT07266181/ICF_002.pdf
  • Informed Consent Form: in Simplified Chinese (2025-10-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT07266181/ICF_003.pdf